CLINICAL TRIAL: NCT04236895
Title: A Glucose Clamp Trial Investigating the Biosimilarity of Gan & Lee Insulin Glargine Injection (Insulin Glargine 100 U/mL) With US and EU Lantus® Comparator Products in Patients With Type 1 Diabetes Mellitus
Brief Title: PK/PD Biosimilarity Study of Gan & Lee Insulin Glargine Injection vs.US & EU Lantus® in Type 1 Diabetes Mellitus Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gan and Lee Pharmaceuticals, USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GL-GLA-CT1002
Record Dates: First submitted 2020-01-15; First posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes; Diabetes Type 1; Type 1; Basal; Insulin; Glargine; T1DM; Diabetes Mellitus; Insulin Dependent Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Insulin Resistance | interventions — gallium nitrate

STUDY DESIGN:
Intervention Model Description: The trial will be a randomized, double-blind, multicenter, single-dose, 3-way crossover, 3-treatment, euglycemic glucose clamp trial in male subjects with type 1 diabetes mellitus
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lantus ® US (Active Comparator): Insulin glargine (Lantus®, product approved and marketed in the USA (US RLD)), 100 U/mL in 3 mL pre-filled pens
  Interventions: Drug: Gan & Lee Insulin Glargine Injection
- Lantus ® EU (Active Comparator): Insulin glargine (Lantus®, product marketed in Germany (EU RP)), 100 U/mL in 3 ml pre-filled pens
  Interventions: Drug: Gan & Lee Insulin Glargine Injection
- Gan & Lee Insulin Glargine (Experimental): Insulin glargine 100 U/mL in 3 mL pre-filled pens
  Interventions: Drug: Gan & Lee Insulin Glargine Injection

INTERVENTIONS:
Drug: Gan & Lee Insulin Glargine Injection — All IMPs will be administered as a 0.5 U/kg single subcutaneous dose by a pre-filled pen.

SUMMARY:
Primary objectives:

To demonstrate biosimilarity with regard to the total and maximum pharmacokinetic exposure during one dosing interval (AUC ins. 0-24h, Cins.

max) of Gan & Lee Insulin Glargine with Lantus® (US RLD / EU RP) in subjects with type 1 diabetes

To demonstrate biosimilarity with regard to the total and maximum pharmacodynamic response during one dosing interval (AUC GIR.0-24h, GIR max) of Gan & Lee Insulin Glargine with Lantus® (US RLD / EU RP) in subjects with type 1 diabetes

Secondary objectives:

To compare the pharmacokinetic and pharmacodynamic properties of Gan & Lee Insulin Glargine and of Lantus® (US RLD / EU RP)

To assess the safety and tolerability of Gan & Lee Insulin Glargine and of Lantus® (US RLD / EU RP)

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent obtained before any trial-related activities. (Trial-related activities are any procedures that would not have been performed during normal management of the subject).
* Male subjects with type 1 diabetes mellitus for at least 12 months prior to screening as diagnosed clinically.
* Age between 18 and 64 years, both inclusive.
* Body Mass Index (BMI) between 18.5 and 29.0 kg/m^2, both inclusive.
* HbA1c <= 9.0%.
* Fasting negative C-peptide (<= 0.30 nmol/L).
* Total insulin dose of < 1.2 (I)U/kg/day.
* Stable insulin regimen for at least 2 months prior to screening (with respect to safety of the subject and scientific integrity of the trial).
* Considered generally healthy (apart from type 1 diabetes mellitus) upon completion of medical history, physical examination, vital signs, ECG and analysis of laboratory safety variables, as judged by the Investigator

Exclusion Criteria:

* Known or suspected hypersensitivity to IMPs or related products
* Previous participation in this trial. Participation is defined as randomized
* Receipt of any medicinal product in clinical development within 30 days or 5 half-lives (whichever is longer) before randomization in this trial
* History of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reaction
* Any history or presence of cancer except basal cell skin cancer or squamous cell skin cancer as judged by the Investigator
* Any history or presence of clinically relevant comorbidity (with the exception of conditions associated with diabetes mellitus), or signs of acute illness, as judged by the Investigator
* Proliferative retinopathy or maculopathy (based on a recent (<1.5 years) ophthalmologic examination) and/or severe neuropathy, in particular autonomic neuropathy, as judged by the Investigator
* Recurrent severe hypoglycemia (more than 1 severe hypoglycemic event during the past 6 months) or hypoglycemic unawareness as judged by the Investigator
* Increased risk of thrombosis, e.g. subjects with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the Investigator
* Significant history of alcoholism or drug abuse as judged by the Investigator or consuming more than 24 grams alcohol/day
* Symptomatic hypotension or supine blood pressure at screening (after resting for at least 5 min in supine position) outside the range of 90-140 mmHg for systolic or greater than 90 mmHg for diastolic pressure
* Heart rate at rest outside the range of 50-90 beats per minute
* Clinically significant abnormal standard 12-lead ECG after 5 minutes resting in supine position at screening, as judged by the Investigator
* A positive result in the alcohol and/or urine drug screen at the screening visit
* Not able or willing to refrain from smoking and use of nicotine substitute products one day before and during the inpatient period
* Positive to the screening test for Hepatitis Bs antigen or Hepatitis C antibodies and/or a positive result to the test for HIV-1/2 antibodies or HIV-1 antigen
* Any medication (prescription and non-prescription drugs) within 14 days before IMP administration, with the exception of occasional use of Paracetamol or NSAIDs
* Blood donation or blood loss of more than 500 mL within the last 3 months
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
* Fertile male with female partner(s) without using a highly effective contraceptive method in combination with spermicide-coated condoms from the first dosing until 1 month after dosing

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 114 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2018-11-28 (Actual)

PRIMARY OUTCOMES:
PK endpoint | Up to 24 hours
  AUCins. 0 - 24h, area under the serum insulin concentration curve from 0 to 24. hours
PK endpoint | Up to 30 hrs
  Cins.max, maximum observed insulin concentration.
PD endpoint | Up to 24 hours
  AUC GIR.0-24h, area under the glucose infusion rate curve from 0 to 24 hours.
PD endpoint | Up to 30 hrs
  GIR max, maximum observed glucose infusion rate

SECONDARY OUTCOMES:
Secondary PK endpoint | Up to 24 hrs
  AUC ins.0-12h, AUC ins.12 - 24h, AUC ins.0 -inf., areas under the serum insulin concentration curve in the indicated time intervals
Secondary PK endpoint | Up to 30 hrs
  tmax.ins, time to maximum observed serum insulin concentration
Exploratory PK endpoint | Up to 30 hrs
  t½, terminal serum elimination half-life calculated as t½=ln2/λz and
Exploratory PK endpoint | Up to 30 hrs
  λz, terminal elimination rate constant
Secondary PD endpoint | Up to 24 hrs
  AUC GIR.0 - 12h, AUC GIR.12 - 24h, areas under the glucose infusion rate curve in the indicated time-intervals
Secondary PD endpoint | Up to 30 hrs
  AUC GIR.0 - last, area under the glucose infusion rate curve from 0 hours until the end of clamp
Secondary PD endpoint | Up to 30 hrs
  t max.GIR, time to maximum glucose infusion rate
Exploratory PD endpoint | Up to 30 hrs
  Duration of action, time until blood glucose levels is consistently above 150 mg/dL
Exploratory PD endpoint | Up to 30 hrs
  Time to onset of action, time from trial product administration until blood glucose concentration has decreased at least 5 mg/dL from baseline, where baseline is defined as the mean of blood glucose levels from - 6 to - 2 minutes before trial product administration as measured by ClampArt.
Safety endpoints | Up to 12 Weeks
  As measured by treatment-emergent adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jia Lu, PhD, Study Director — Gan & Lee Pharmaceuticals, USA; Leona Plum - Mörschel, MD, PD, Principal Investigator — Profil Mainz GmbH & Co KG
Locations (2):
- Germany (2):
  - Profil Mainz GmbH & Co. KG, Mainz
  - Profil Institut für Stoffwechselforschung GmbH, Neuss

REFERENCES:
- [Derived] Chen W, Lu J, Plum-Morschel L, Andersen G, Zijlstra E, He A, Xie T, Li L, Hao C, Gan Z, Heise T. Pharmacokinetic and pharmacodynamic bioequivalence of Gan & Lee insulin analogues aspart (rapilin(R)), lispro (prandilin(R)) and glargine (basalin(R)) with EU- und US-sourced reference insulins. Diabetes Obes Metab. 2023 Dec;25(12):3817-3825. doi: 10.1111/dom.15281. Epub 2023 Sep 21. PMID 37735841